CLINICAL TRIAL: NCT01852903
Title: A Randomized, Double-blind, Placebo-controlled Crossover Study Comparing the Bioavailability of Two Forms of Vitamin C in Plasma and Leukocytes Over 24 Hours.
Brief Title: Comparative Bioavailability of Two Forms of Vitamin C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NBTY, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry); Moyad, Mark MD MPH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11CIHE
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Bioavailability
Keywords: vitamin C; calcium ascorbate; ascorbic acid; bioavailability
MeSH Terms: interventions — calcium ascorbate; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- calcium ascorbate (Experimental)
  Interventions: Dietary Supplement: calcium ascorbate
- ascorbic acid (Active Comparator)
  Interventions: Dietary Supplement: ascorbic acid
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: calcium ascorbate
  Other Names: vitamin C
  Arms: calcium ascorbate
Dietary Supplement: ascorbic acid
  Other Names: vitamin C
  Arms: ascorbic acid
Other: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to compare levels of vitamin C in the blood over the 24 hour period following a single 1000 mg dose of vitamin C from ascorbic acid, calcium ascorbate and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by laboratory results and medical history
* Females not of child bearing potential
* BMI 18-30 kg/m2
* Agrees to consume a low vitamin C diet
* Non-smoker or ex-smoker >1 year

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during the trial
* Alcohol >2 drinks per day; alcohol or drug abuse within the past year
* Cardiac conditions
* Duodenal ulcer or gastric ulcer, gastritis, hiatus hernia, or gastroesophageal reflux disease (GERD) within past 3 months
* History irritable bowel syndrome, malabsorption or significant GI disease
* History of kidney stones
* Use of medications known to interact with vitamin C
* Use of supplements containing vitamin C
* Use of anticoagulants (warfarin), barbiturates, tetracycline antibiotics, beta-blockers, cyclosporine, prednisone, tricyclic antidepressants, diuretics and nitrate medications
* History of or current diagnosis of cancer
* Uncontrolled hypertension
* History of diabetes, renal disease and/or liver disease
* Unstable psychiatric disorder
* History of or current immunocompromise
* History of hemochromatosis or hemoglobinopathies
* Participation in a clinical research trial <30 days
* Use of acute medication w/in 72 hours of intervention
* Unstable medications <90 days
* Abnormal liver function
* Serum creatinine > 1.5 x upper limit of normal (ULN)
* Anemia of any etiology
* Blood donation w/in the last 2 months
* Allergy or sensitivity to test articles, foods or beverages provided during the study
* Cognitive impairment and/or unable to give informed consent

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Plasma and leukocyte vitamin C concentration | 0, 2, 4, 8 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dale R Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc, London, Ontario, Canada

REFERENCES:
- [Derived] Mitmesser SH, Ye Q, Evans M, Combs M. Determination of plasma and leukocyte vitamin C concentrations in a randomized, double-blind, placebo-controlled trial with Ester-C((R)). Springerplus. 2016 Jul 25;5(1):1161. doi: 10.1186/s40064-016-2605-7. eCollection 2016. PMID 27512620